CLINICAL TRIAL: NCT02146547
Title: European Long-acting Antipsychotics in Schizophrenia Trial
Acronym: EULAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Rene Kahn, Professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABR49490
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Schizophrenia
Keywords: depot, oral, antipsychotics, paliperidone, aripiprazole
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- aripiprazole oral (Active Comparator): the recommended starting dose for aripiprazole is 10 or 15 mg/day with a maintenance dose of 15 mg/day administered on a once-a-day schedule without regard to meals.Aripiprazole is effective in a dose range of 10 to 30 mg/day.
  Interventions: Drug: Aripiprazole
- Aripiprazole depot (Active Comparator): The recommended starting and maintenance dose of aripiprazole depot is 400 mg. Titration of the dose of this medicinal product is not required. It should be administered once monthly as a single injection (no sooner than 26 days after the previous injection).
  After the first injection, treatment with 10 mg to 20 mg oral aripiprazole should be continued for 14 consecutive days to maintain therapeutic aripiprazole concentrations during initiation of therapy.
  If there are adverse reactions with the 400 mg dosage, reduction of the dose to 300 mg once monthly should be considered.
  Interventions: Drug: Aripiprazole depot
- Paliperidone (Active Comparator): The recommended dose of paliperidone for the treatment of schizophrenia is 6 mg once daily, administered in the morning. Initial dose titration is not required. Some patients may benefit from lower or higher doses within the recommended range of 3 mg to 12 mg once daily. Dosage adjustment, if indicated, should occur only after clinical reassessment. When dose increases are indicated, increments of 3 mg/day are recommended and generally should occur at intervals of more than 5 days.
  Interventions: Drug: Paliperidone
- Paliperidone palmitate (Active Comparator): The first two administrations of paliperidone palmitate (150 mg at visit 3 and 100 mg one week later) need to be administered deep into the deltoid muscle in order to attain therapeutic concentrations rapidly. No oral supplementation with paliperidone is needed. Following the second dose, monthly maintenance doses can be administered in either the deltoid or gluteal muscle. The recommended monthly maintenance dose is 75 mg, although some patients may benefit from lower doses within the recommended range of 25 to 150 mg based on individual patient tolerability and/or efficacy.
  Interventions: Drug: Paliperidone palmitate

INTERVENTIONS:
Drug: Aripiprazole — Administration in once-a-day schedule without regard to meals.
  Other Names: Abilify
  Arms: aripiprazole oral
Drug: Aripiprazole depot — Abilify Maintena is an intramuscular (IM) depot formulation of oral aripiprazole. It provides the efficacy and safety profile of oral aripiprazole in a once-monthly injection.
  Other Names: Abilify maintena
  Arms: Aripiprazole depot
Drug: Paliperidone — Administration once a day orally standardised in relation to food intake.
  Other Names: Invega
  Arms: Paliperidone
Drug: Paliperidone palmitate — In selected patients with schizophrenia and previous responsiveness to oral paliperidone or risperidone, Xeplion may be used without prior stabilization with oral treatment if psychotic symptoms are mild to moderate and a long-acting injectable is needed.
  Other Names: Xeplion
  Arms: Paliperidone palmitate

SUMMARY:
Schizophrenia is a chronic psychiatric illness with periods of remission and relapse. Patients vary in the frequency and severity of relapse, time until relapse and time in remission. Discontinuation of antipsychotic medication is by far the most important reason for relapse. A possible method to optimize medication adherence is to treat patients with long-term, depot medication rather than oral medication. However, despite its apparent "common sense" this approach has neither been universally accepted by practicing psychiatrists nor unequivocally demonstrated in clinical trials. Therefore, in this study we aim to investigate possible advantages of depot medication over oral antipsychotics in an independently designed and conducted, randomized, pragmatic trial.

DETAILED DESCRIPTION:
It remains unclear if depot medication can reduce relapse rates and improve clinical outcome when offered to all patients in need of continuation treatment with antipsychotics. Before we can conclude whether or not all schizophrenia patients could benefit from a switch to depot formulations, several questions remain to be answered. Is depot medication associated with better continuation rates and outcome? How are depot medications tolerated as compared to oral medication? In order to clarify these important issues we aim to perform a large multi-center trial in which schizophrenia patients in need of continuous treatment who are randomized 1:1:1:1 to two different depot preparations or to two different oral medications.

In this pragmatic, randomized, open label, multicenter, multinational comparative trial, schizophrenic patients aged 18 years or older, having experienced the first psychosis between 6 months and 7 years ago,with an indication (patient or physician initiated) to receive medication or to switch to another antipsychotic drug, will enter the study.

The study duration will be one month for the medication switch and then a follow-up of 18 months. Patients having refused to take part in the study will be asked to give consent and participate in a naturalistic follow-up, during which they will be followed with the Clinical Global Impression list (CGI) as closely related to the study schedule as possible, unless they also refuse this.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia as defined by DSM-IV-R (Diagnostic and Statistical Manual) as determined by the M.I.N.I.plus
2. Age 18 or older.
3. 3. The first psychosis occurred at least 6 months and no more than 7 years ago.*
4. If patients are using an antipsychotic drug, a medication switch is currently under consideration.
5. Capable of providing written informed consent

   * Time of first psychosis is defined as the first contact with a health care professional in relation to psychotic symptoms.

Exclusion Criteria:

1. Intolerance / hypersensitivity to both* of the drugs (including active substances, metabolites and excipients) in this study including oral paliperidone and aripiprazole and/or hypersensitivity to risperidone.
2. Pregnancy or lactation.
3. Patients who are currently using clozapine.
4. Patients who do not fully comprehend the purpose or are not competent to make a rational decision whether or not to participate.
5. Patients with a documented history of intolerance to both* of the study medications and/or a documented history of non-response to a treatment with both* study drugs of at least 6 weeks within the registered dose range.7. Patients who have been treated with an investigational drug within 30 days prior to screening.

8. Simultaneous participation in another intervention study (neither medication or psychosocial intervention).

* If intolerance/hypersensitivity or non-response in the past to one of the compounds is documented, the patient can still participate; however, randomization will take place by blocking that specific compound. That is, the patient will be randomized on either the oral or the depot arm of the other compound. This procedure of blocking one compound is also accepted for patients who have experienced too many side effects to one of the compounds in the past, as documented in the patient's medical record. The decision to block that specific compound for randomization in these cases is up to the discretion of the treating physician who will carefully balance this decision and clearly document it in the medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
All cause discontinuation rates | 18 months
  Compare all cause discontinuation rates in patients with schizophrenia randomized to oral antipsychotic medications (i.e., aripiprazole or paliperidone) versus depot antipsychotic medications (i.e., paliperidone palmitate or aripiprazole depot).
  Discontinuation consist of (multiple options are possible):
  * the allocated treatment is stopped or used at doses outside the allowed range.
  * medication is switched or augmented with another antipsychotic after visit 4 for more than 1 month continuously or for more than 3 months cumulative over the 18 months of the trial.
  * a patient misses a monthly visit and does not show up after reminding him
  * patient withdraws consent for the study.
  * clinician decision to withdraw the patient.

SECONDARY OUTCOMES:
Subjective Wellbeing under Neuroleptics | 18 months
  Change from baseline in Subjective Wellbeing under Neuroleptics
EuroQoL quality of life scale | 18 months
  Change from baseline in EuroQoL quality of life scale
Side effects assessment | 18 months
  Change from baseline in SMARTS (Systematic Monitoring of Adverse events Related to TreatmentS) and the Abnormal and Involuntary Movement Scale.
Assessment of cognitive functioning | 18 months
  Compare the combined oral medication group with the combined depot treatment arms regarding cognitive functioning
Assessment of Positive and Negative Symptom Scale | 18 months
  Compare the combined oral medication group with the combined depot treatment arms regarding changes in different dimensions of psychopathology of schizophrenia
Assessment of Personal and Social Performance Scale | 18 months
  Compare the combined oral medication group with the combined depot
Change from baseline of Personal and Social Performance Scale | Baseline until 18 months
  Compare the combined oral medication group with the combined depot

OTHER OUTCOMES:
Comparison between depot arms and the oral treatment arms on the one side | 18 months
  The comparisons will also be made between the depot arms and the oral treatment arms on the one side and the patients who are followed up naturalistically.Depot arms are compared regarding augmentation with oral antipsychotics after visit 4.
Treatment success regarding outcomes in patients who have not given consent for the main trial | up to 18 months
  compare treatment success regarding the outcomes mentioned above to those achieved in a group of patients who did not agree to participate in the trial but could be followed up with the CGI.
Compare side effects between combined oral medication groups & combined depot treatment | 18 months
  Compare side effects and general wellbeing under antipsychotic medication between the combined oral medication groups with the combined depot treatment arms.
Immune parameters | 18 months
  Associations between immune parameters on the one hand, and primary as well as secondary outcome measures on the other.

CONTACTS AND LOCATIONS:
Overall Officials: Rene S Kahn, professor, Principal Investigator — UMC Utrecht; Wolfgang Fleischhacker, professor, Principal Investigator — Department of Biological Psychiatry, Innsbruck University Clinics; Michael Davidson, professor, Principal Investigator — Department of Psychiatry, Sackler Faculty of Medicine, Tel Aviv University, Israel
Locations (49):
- Austria (2):
  - Department of Biological Psychiatry, Innsbruck University Clinics, Innsbruck, Anichstrasse 35
  - Psychosoziale Dienste, Vienna, Modecenterstraße
- Belgium (2):
  - ZNA, department of Psychiatry, locatie Stuivenberg, Antwerp, Lange Beeldekensstraat 267
  - Psychiatrisch Ziekenhuis Duffel, Antwerp, Stationsstraat 22C
- University Hospital of Neurology and Psychiatry 'St. Naum' 1, Sofia, Louben Roussev Str., Bulgaria
- Czechia (3):
  - Psychiatrická klinika LF UK, Hradec Králové, Fakultní Nemocnice
  - Dr. Ustohal, Brno
  - Dr. Mohr, Prague
- Center for Neuropsychiatric Research, Glostrup Municipality, Ndr. Ringvej, Denmark
- Germany (4):
  - Klinik und Poliklinik für Psychiatrie und Psychotherapie der Heinrich-Heine-Universität, Düsseldorf, Bergische Landstraße 2
  - Technische Universität München (TUM, München, Ismaningerstrasse 22
  - Klinik für Psychiatrie, Psychotherapie und Psychosomatik der Martin-Luther-Universität, Halle, Julius-Kühn-Straße 7
  - Department of Psychiatry and Psychotherapy, München, Nussbaumstrasse 7
- National and Kapodistrian University of Athens Medical School, Eginition Hospital, Athens, Greece
- Hungary (2):
  - Dr. Csekey, Balassagyarmat
  - Department of Psychiatry and Psychotherapy, Semmelweis University, Budapest
- Israel (6):
  - Abravanel Mental Health Center, Bat Yam
  - Be'er-Ness Mental Health Center, Be’er Ya‘aqov
  - The Jerusalem Mental Health Center, Jerusalem
  - Lev-Hasharon Medical Center for Mental Health, Pardesiyya
  - Geha Medical Health Center, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - Department of Psychiatry, University of Naples SUN, Naples, Largo Madonna Delle Grazie 1
  - Università degli Studi di Torino. Dipartimento di Neuroscienze, Turin, Sezione Di Psichiatriavia Cherasco, 11
  - Servizio Psichiatrico Universitario di Diagnosi e Cura. Presidio Ospedaliero "San Salvatore" Università degli Studi dell'Aquila., L’Aquila
- University Medical Center, Utrecht, Netherlands
- Norway (3):
  - Helse Bergen HF Haukeland University Hospital, Division of Psychiatry, Bergen
  - Stavanger University Hospital, Stavanger
  - St Olavs Hospital avd Østmarka / INM NTNU, Trondheim
- Poland (2):
  - Instytut psychiatrii i neurologii, Warsaw, Sobieskiego 9
  - II Klinika Psychiatrii Uniwersytet Medyczny w Lublinie, Lublin, Ul. Głuska 1
- Romania (6):
  - Spitalul Clinic Judetean de Urgenta Arad - Clinica de Psihiatrie, Arad
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia", Bucharest
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia, Bucharest
  - Spitalul de Psihiatrie si pentru Masuri de Siguranta, Sapoca, Buzau, Buzău
  - Spitalul Clinic de Neuropsihiatrie Craiova, Craiova
  - Sitalul Clinic Judetean Mures, Targu Mureş
- Spain (4):
  - Hospital Clínic de Barcelona. Unidad de Esquizofrenia, Barcelona, C/Villarroel, 170. Escalera12, Planta 0
  - Hospital Universitario Marqués de Valdecilla, Servicio de Psiquiatría, Santander, Cantabria
  - Facultad de Medicina Center, Oviedo, Julián Clavería S/n
  - Child and Adolescent Psychiatry Department. Hospital General Universitario Gregorio Marañón. Servicio Madrileño de Salud, Madrid
- United Kingdom (8):
  - West London Mental Health Trust. East Recovery Team, London, Avenue House 43-47 Avenue Road
  - Greater Manchester West Mental Health NHS Foundation Trust, Manchester, Crowell House, Cromwell Road
  - Edmund Ward, St Martins Hospital Littlebourne Road Canterbury, Kent
  - Imperial College, Centre for Mental Health, Faculty of Medicine,, London
  - Tees, Ask and Wearvalleys, Middlesbrough
  - Northumberland, Newcastle
  - Oxford Health NHS Foundation Trust, Oxford
  - Surrey and Borders Partnership NHS Foundation Trust, Surrey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mortazavi M, Aminifarsani Z, Rossum IW, Kahn RS, Fleischhacker WW, Davidson M, Weiser M, Siskind D, Leucht S; EULAST Study Group; Hasan A, Wagner E. Impact of Long-Acting Injectable Versus Oral Antipsychotic Treatment on All-Cause Discontinuation Risk in People with Early Phase Schizophrenia and Comorbid Substance Use Disorder: A Secondary Analysis of the EULAST Randomized Trial. CNS Drugs. 2026 Jan;40(1):99-109. doi: 10.1007/s40263-025-01225-0. Epub 2025 Sep 11. PMID 40932600
- [Derived] Winter-van Rossum I, Weiser M, Galderisi S, Leucht S, Bitter I, Glenthoj B, Hasan A, Luykx J, Kupchik M, Psota G, Rocca P, Stefanis N, Teitelbaum A, Bar Haim M, Leucht C, Kemmler G, Schurr T; EULAST Study Group; Davidson M, Kahn RS, Fleischhacker WW. Efficacy of oral versus long-acting antipsychotic treatment in patients with early-phase schizophrenia in Europe and Israel: a large-scale, open-label, randomised trial (EULAST). Lancet Psychiatry. 2023 Mar;10(3):197-208. doi: 10.1016/S2215-0366(23)00005-6. Epub 2023 Jan 27. PMID 36716759